CLINICAL TRIAL: NCT07312058
Title: Long-term Evaluation of Fertility Preservation Options in Women in Cancer Remission or Haematological Pathology
Acronym: FERT-ISSUES
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2025_843_0156
Record Dates: First submitted 2025-11-17; First posted 2025-12-31 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Fertility Preservation; Cancer Remission; Reproductive Outcomes; Reproductive Health; Oncology; Fertility Counseling; Assisted Reproductive Technology; Psychological Impact; Fertility Observatory; Patient Follow-up; Female Cancer Survivors; Fertility Preservation Techniques; Live Birth Rate
Keywords: Fertility preservation; Cancer remission; Reproductive outcomes; Reproductive health; Oncology; Fertility counseling; Assisted reproductive technology; Psychological impact; Fertility observatory; Patient follow-up; Female cancer survivors; Fertility preservation techniques; Live birth rate
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cancer treatments, despite their increasing effectiveness, carry a significant risk of gamete toxicity.

Women of reproductive age are commonly offered fertility preservation (FP) before starting their treatment.

However, few studies have analyzed the long-term reproductive outcomes of these interventions, nor how patients ultimately use or do not use the FP options once in remission.

This project aims to better understand the effectiveness, utilization, and psychological impacts of these strategies.

This work is part of an effort to understand and evaluate fertility preservation practices implemented for women of reproductive age undergoing cancer treatment at the Amiens-Picardie University Hospital (CHU).

Its objective is to document patient pathways, clinical decisions, techniques employed, and reproductive outcomes observed after remission, in order to identify potential areas for improvement in the support and follow-up of these patients, thereby enhancing the overall quality and coordination of care.

This work is conducted alongside the development of a fertility observatory at the Department of Medicine and Reproductive Biology, CHU Amiens-Picardie.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Aged between 18 and 47 years
* Diagnosed with cancer or hematological disorders requiring potentially gonadotoxic treatment
* Having undergone a medical fertility preservation consultation
* Followed at Amiens Picardie University Hospital (CHU Amiens Picardie) in the department of Reproductive Medicine
* Currently in remission
* Having expressed non-opposition to participation in the study

Exclusion Criteria:

* Absence of remission
* Patients deprived of liberty by administrative or judicial decision, or placed under legal protection (guardianship or curators)
* Decline to participate in the study

Ages: 18 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — * Women
  * Aged between 18 and 47 years
  * Diagnosed with cancer or hematological disorders requiring potentially gonadotoxic treatment
Study Population: Patients are recruited during follow-up consultations as part of the establishment of a fertility observatory within the Department of Medicine and Reproductive Biology at CHU Amiens Picardie
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2025-12-17 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of an identifiable reproductive outcome | 1 year
  Identifiable reproductive outcome are Spontaneous pregnancy, Use of preserved gametes or ovarian tissue (whether or not resulting in pregnancy), Use of donor oocytes, Discontinuation of the parenthood project

SECONDARY OUTCOMES:
Type of fertility preservation method performed | 1 year
Time interval (in months) between diagnosis and fertility preservation | 1 year
Correlation between Age and occurance of an identifiable reproductive outcome | 1 year
  Identifiable reproductive outcome are Spontaneous pregnancy, Use of preserved gametes or ovarian tissue (whether or not resulting in pregnancy), Use of donor oocytes, Discontinuation of the parenthood project
Time interval (in months) between fertility preservation and initiation of potentially gonadotoxic treatment | 1 year
Number of type of cancer associated with identifiable reproductive outcome | 1 year
  Identifiable reproductive outcome are Spontaneous pregnancy, Use of preserved gametes or ovarian tissue (whether or not resulting in pregnancy), Use of donor oocytes, Discontinuation of the parenthood project
Correlation between type of treatment and occurence of an identifiable reproductive outcome | 1 year
  Identifiable reproductive outcome are Spontaneous pregnancy, Use of preserved gametes or ovarian tissue (whether or not resulting in pregnancy), Use of donor oocytes, Discontinuation of the parenthood project
Correlation between family status and occurence of an identifiable reproductive outcome | 1 year
  Identifiable reproductive outcome are Spontaneous pregnancy, Use of preserved gametes or ovarian tissue (whether or not resulting in pregnancy), Use of donor oocytes, Discontinuation of the parenthood project
Time interval (in months) between completion of treatment and pregnancy attempt (spontaneous or medically assisted) | 1 year
Actual utilization rate of preserved material | 1 year
Success rate of reuse attempts | 1 year
Proportion of patients who ultimately did not pursue parenthood | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No